CLINICAL TRIAL: NCT06729164
Title: Randomized Controlled Trial: Strategic and Interactive Signing Instruction
Brief Title: Strategic and Interactive Signing Instruction Experiment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 451965; 1R21DC021024-01A1 (NIH)
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Sign Language Skills; Teacher Practice
Keywords: Deaf; Sign language; Instruction; Intervention
MeSH Terms: conditions — Sign Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RCT - Experimental (Experimental): This RCT study involves teachers divided into an experimental group and a control group. Teachers in the experimental group will receive SISI training to support the sign language development of deaf children, while those in the control group will continue with "business-as-usual" teaching methods. Pre- and post-assessments will be conducted for all deaf children at the beginning and end of the school year.
  Interventions: Behavioral: Strategic and Interactive Signing Instruction
- Quasi-Experimental Study - Control (Placebo Comparator): This quasi-experimental study involves teachers divided into an experimental group and a control group. Teachers in the experimental group will receive SISI training to support the sign language development of deaf children, while those in the control group will continue with "business-as-usual" teaching methods. Pre- and post-assessments will be conducted for all deaf children at the beginning and end of the school year.
  Interventions: Behavioral: Business-As-Usual Instruction

INTERVENTIONS:
Behavioral: Strategic and Interactive Signing Instruction — Evidence-based instructional methods guided by cognitive, sociocultural, and linguistic theories that are applied to interventions supporting sign language development among deaf children.
  Arms: RCT - Experimental
Behavioral: Business-As-Usual Instruction — Teachers will teach business-as-usual without the inclusion of SISI.
  Arms: Quasi-Experimental Study - Control

SUMMARY:
This RCT study involves teachers divided into an experimental group and a control group. Teachers in the experimental group will receive SISI training to support the sign language development of deaf children, while those in the control group will continue with "business-as-usual" teaching methods. Pre- and post-assessments will be conducted for all deaf children at the beginning and end of the school year.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) examines the effects of the Strategic and Interactive Signing Instruction (SISI) intervention on deaf children's expressive language development in signing (primary) and writing (secondary). The study compares two groups - an intervention group implementing SISI and a control group continuing their usual instructional routines without the intervention.

The intervention group will include approximately 10 teachers, each working with 5-7 deaf children. These classrooms will implement the SISI intervention, which provides structured, language-centered supports designed to strengthen children's signing through explicit modeling, guided practice, and discourse-focused intervention routines. Schools that participated in the 2024-2025 nationwide pre/post study will be included in the intervention group for 2025-2026 if they choose to continue.

The control group will likewise include approximately 10 teachers with 5-7 Deaf children each. These classrooms will continue with their standard practices without the SISI intervention. Schools newly joining the project in 2025-2026 will be assigned to this group.

Child language data will be collected twice - fall 2025 (pre-test) and spring 2026 (post-test). Deaf children will complete three expressive language prompts representing major discourse types: personal narrative, informational report, and persuasive discourse. Their signed and written compositions will be analyzed using rubrics adapted from the National Assessment of Educational Progress (NAEP), focusing on growth in discourse-level skills.

The study hypothesizes that deaf children in the intervention group will show greater gains in expressive signing and writing than their peers in the control group. This hypothesis reflects the expectation that a systematic, discourse-oriented language intervention offers stronger support for language development than typical intervention routines.

This research aims to contribute to the evidence base on interventions that support deaf children's expressive language development. By examining child-level language outcomes from a discourse-focused intervention, the study will advance understanding of how structured language support can strengthen signing and writing development for deaf children.

ELIGIBILITY:
Inclusion Criteria:

* Deaf children in educational programs (aged 4-12)
* Teachers of the deaf working with deaf children

Exclusion Criteria:

* Non-deaf children
* Non teachers of the deaf

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Sign Language Skills | From enrollment to the end of treatment 9 academic months later.
  Student data will be analyzed using rubrics adapted from the National Assessment of Educational Progress (NAEP) standardized writing assessments.
Teacher Practice | From enrollment to the end of treatment 9 academic months later.
  The SISI Fidelity Tool, grounded in existing literature on evidence-based instructional methods, will be used to evaluate teachers' instructional practices.

SECONDARY OUTCOMES:
Written Language Skills | From enrollment to the end of treatment 9 academic months later.
  Student data will be analyzed using rubrics adapted from the National Assessment of Educational Progress (NAEP) standardized writing assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Leala Holcomb, PhD, Principal Investigator — Center of Deafness
Locations (1):
- University of Tennessee, Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Under a data-sharing agreement that is in compliance with the internal policy at UTK, non-identifying data can be shared with other researchers for a minimum of 10 years on the University of Tennessee Research and Creative Exchange (TRACE). The raw data consists of videos of teachers, which will not be shared to maintain confidentiality. The processed data will be in the form of percentages for individual teachers across an academic year documented in a .csv file (Excel). Center for Open Science Foundation (OSF) is a free and open source project management tool that supports researchers throughout their entire project lifecycle. OSF also allows people to locate this data through project names, author names, and study keywords.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December, 2026 to December, 2036
Access Criteria: Researchers may contact the principal investigator for additional supporting information not available on OSF.

REFERENCES:
- [Background] Holcomb L, Eberwein AA. Teacher reports of ASL literacy instruction in deaf education. J Deaf Stud Deaf Educ. 2025 Oct 7:enaf060. doi: 10.1093/jdsade/enaf060. Online ahead of print. PMID 41055392
- [Background] Holcomb L. Exploring signed literacy in elementary deaf students through evidence-based instructional methods. Sign Language Studies. 2024; 24(4):843-882.
- See also: Website about the research project — https://cehhs.utk.edu/tpte/asl-literacy-instruction-in-deaf-education/
- Available data/document: The study's relevant instructional context measures. Supporting materials include the assessment instrument, protocols, etc.: Open Science Framework — https://osf.io/eq5s8/overview